CLINICAL TRIAL: NCT07291180
Title: A Feasibility Study of Mass-Based Response Drug Screening to Guide Personalized Hyperthermic Intraperitoneal Chemotherapy for High-Grade Appendiceal and Colorectal Adenocarcinoma With Peritoneal Metastasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Travera Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000038133
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Appendiceal Cancer; Colorectal Adenocarcinoma; Peritoneal Metastases
Keywords: Appendiceal Cancer; Colorectal Adenocarcinoma; Peritoneal Metastases; Iterative Hyperthermic Intraperitoneal Chemotherapy (IHIPEC)
MeSH Terms: conditions — Appendiceal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with peritoneal metastasis from high-grade appendiceal and colorectal adenocarcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MRT (Experimental): Participants with high-grade appendiceal and colorectal peritoneal metastasis will receive MRT to select and deliver personalized HIPEC regimens to participants undergoing IHIPEC
  Interventions: Device: Mass-based response testing (MRT)

INTERVENTIONS:
Device: Mass-based response testing (MRT) — Travera has developed a clinical workflow that combines single-cell mass measurements with inline brightfield imaging and machine-learning based image classification to perform mass-based response testing (MRT) directly on live tumor cells collected from patients. MRT enables tumor cells across a wide range tissue sample formats to be dosed with a panel of drugs in vitro, agnostic to malignancy or drug mechanism.

SUMMARY:
This study will evaluate the role of mass-based response testing (MRT) to select and deliver personalized hyperthermic intraperitoneal chemotherapy (HIPEC) regimens to patients with peritoneal metastasis (PM) from high-grade appendiceal adenocarcinomas (HGAA) and colorectal cancer (CRC).

DETAILED DESCRIPTION:
Patients with peritoneal metastases from colorectal and appendix cancer are treated with cytoreductive surgery and HIPEC. However, several patients are considered unresectable due to the inability to remove all the cancer safely. Repeated (Iterative) intra-peritoneal chemotherapy delivered via HIPEC laparoscopically has been shown to have favorable outcomes with a potential increase in sensitivity to immunotherapy . Such procedures often use chemotherapy that is not tailored to the patients cancer.

In this study, patients with unresectable colorectal and appendiceal peritoneal metastases will undergo MRT on tissue biopsies to determine optimal chemotherapy regimen to be delivered intraperitoneally. For patients with unresectable disease, iterative HIPEC (IHIPEC) will be administered starting three weeks after the laparoscopy. (IHIPEC refers to HIPEC followed by systemic chemotherapy repeated 3 times with approximately 6 weeks in between each HIPEC.)

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed peritoneal metastases with primary diagnosis of AJCC 8th Edition Stage IV

  1. Appendiceal adenocarcinoma (moderately/poorly differentiated, and/or signet ring cell tumors)
  2. Colorectal adenocarcinoma
  3. Suspected colon, small bowel, or appendiceal adenocarcinoma in setting of unknown primary
* Limited or no extraperitoneal metastases (any of the below)

  a) Any extraperitoneal metastases must be limited, stable and treatable
* Has adequate organ function, as described below; all screening laboratory tests should be performed within 30 days prior to the first HIPEC
* Expected survival at the time of first HIPEC is greater than 3 months
* Exhibits unresectable disease (bowel or mesenteric involvement) or PCI > 19

Demographics

* Adult patient at least 18 years of age at the time of signing informed consent and less than 81 years of age at the time of signing informed consent.
* Has an ECOG performance status score of 0-2.

Male Participants

* A male participant must agree to use contraception (barrier birth control, abstinence) during the treatment period and for at least 95 days following completion, corresponding to time needed to eliminate any study intervention(s), and refrain from donating sperm during this period.

Female Participants

* A female participant of childbearing age is eligible to participate if she is not pregnant, not breastfeeding, and agrees to use contraception (hormonal, barrier birth control, or abstinence). Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.

Informed Consent

* The participant (or legally acceptable representative if applicable) provides written informed consent for the study. The participant may also provide consent for FBR. However, the participant may participate in the main study without participating in FBR.

Alternative Eligibility

* In addition to the criteria above, if a patient has undergone less than 8 rounds of chemotherapy at another institution (prior to initial diagnostic laparoscopy) and has not undergone radiation, ablative procedures, or cytoreductive surgery, then they are still eligible to enter the study at the second diagnostic laparoscopy step

Exclusion Criteria:

* Has a positive urine pregnancy test within 3 days prior to randomization or treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has a known allergy to medications used in this study. Note: In the event that 3 days have elapsed between the screening pregnancy test and the first dose of study intervention, another pregnancy test (urine or serum) must be performed and must be negative for the participant to start receiving study medication.
* Has hypoxia as defined by pulse oximeter reading <92% at rest or requires intermittent or chronic supplemental oxygen.
* No concurrent malignancy that may interfere with the study aims at the discretion of the investigator.

Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

* Has known significant extraperitoneal metastasis.
* Has creatine clearance <60 mL/m^2 per the Cockcroft-Gault formula
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from treatment initiation, or New York Heart Association Class III or IV congestive heart failure. Medially controlled arrhythmia stable on medication is permitted.
* Has poorly controlled hypertension defined as SBP ≥150mmHg and/or DBP ≥90mmHg.
* Has moderate to severe hepatic impairment (Child-Pugh B or C).
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (severe dysphasia, bowel obstruction, malabsorption).
* Has progressive disease following the first 3 months of systemic chemotherapy prior to HIPEC who is not in a stable condition to continue with the trial.

Prior/Concomitant Therapy

* Has received radiation, ablative procedures, cytoreductive surgery, or systemic therapy including chemotherapy to treat metastatic disease within 3 months of initial laparoscopy.

Diagnostic Assessments

* Has an active infection requiring systemic therapy.
* Has a known active TB/ COVID infection.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study intervention.
* Has a known history of poorly controlled HIV infection despite anti-retroviral therapy.
* Has a known history of HBV (defined as HBsAg reactive) or known active HCV (defined as HCV RNA [qualitative] is detected) infection that is poorly controlled.

Note: Testing for HBV and HCV is only required if mandated by the local health authority.

Other Exclusions

* Inability to receive chemotherapy due to medical/insurance reasons.
* Requires emergency surgery due to bleeding, perforation, or obstruction.
* Has undergone previous iterative intraperitoneal therapy.
* Has contraindication to chemotherapy of choice.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of performing MRT to select and deliver personalized HIPEC | at end of study, up to 12 months
  Feasibility is defined as the percentage of treatment naïve and pretreated patients who successfully receive drug screening results within one week of tissue sampling from at least one peritoneal biopsy. This means that the test has enough tumor cell viability and purity to come back with specific results indicating sensitivities of HIPEC drugs and does not give an inconclusive result (due to insufficient tissue sample).

SECONDARY OUTCOMES:
Concordance of MRT Results | at end of study, up to 12 months
  Defined as the percentage of patients who receive identical HIPEC recommendations (reflecting the best response to MRT) in both rounds of testing. Concordance will only be evaluated for the subset of patients who have received two biopsies and Travera screenings.
One Year Overall Survival (OS) | up to 12 months
  Overall survival of patients will be measured from two time points: From the diagnosis of peritoneal metastasis to death from any cause at the end of follow-up (1 year).
  From the first HIPEC procedure to death from any cause at the end of follow-up (1 year).
Percentage of participants with Perioperative and Postoperative Complications | up to 12 months
  Percentage of participants that experienced any perioperative or postoperative complications will be graded using the CTCAE version 5. Complications will be noted during hospitalization or within 30 days of each HIPEC procedure, and incidence will be measured separately for patients undergoing IHIPEC.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC-QLQ-C30) mean score | every 3 months post last IHIPEC, up to 12 months
  A tool used to assess the quality of life in cancer patients. It contains 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single symptom items (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact) 10. It is scored on a 4-point scale (1 = not at all, 2 = a little, 3 = quite a bit, 4 = very much). The EORTC QLQ-C30 instrument also contains 1 global health status/QoL scale that uses a 7-point scale scoring with anchors (1 = very poor and 7 = excellent).
Change in Comprehensive Score for Financial Toxicity (COST) | every 3 months post last IHIPEC, up to 12 months
  The COST is a standardized instrument for use as a measure of financial toxicity. The COST questionnaire is a patient-friendly tool that has demonstrated reliability, validity, and internal consistency. It has demonstrated an association with health-related quality of life (HRQOL). It contains 12 brief statements about the financial burden, cost, resources, and concerns related to them. It is scored by the patients on a 5-point scale (0=not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4=very much). A composite score is then calculated, with a lower score indicating financial toxicity.
Change in Peritoneal Regression Grading Score (PRGS) | at first IHIPEC post biopsy to last IHIPEC received, up to 12 months
  PRGS is a scoring system used to assess tumor regression in biopsies from patients with peritoneal metastasis undergoing therapy. Peritoneal punch biopsies will be collected from all four abdominal quadrants at the start of each IHIPEC procedure. The attending pathologist will evaluate each biopsy and assign a grade, ranging from 1 (indicating a complete response) to 4 (indicating no response). These individual scores will then be averaged to calculate the overall PRGS score. The change in PRGS is defined as the difference in PRGS between the first and last IHIPEC procedure that a patient receives.
Change in Peritoneal Cancer Index (PCI) Score | during each diagnostic laparoscopy at approximately month 1 and month 6
  The change in PCI score will only be measured for patients undergoing IHIPEC. The PCI is a scoring system used to quantify the extent of peritoneal carcinomatosis. The abdomen is divided into 13 regions and assigned a score ranging from 0 to 3 based on presence and size of peritoneal tumor implants in each region. This score can range from 0 (no evidence of disease) to 39 (extensive disease). PCI scores will be assessed and recorded by the attending physician following peritoneal cavity exploration before each IHIPEC procedure. The change in PCI score is defined as the difference in PCI between the first and last IHIPEC procedure that a patient receives.
Complete Cytoreduction Rate | during each IHIPEC cycle, up to 12 months
  The complete cytoreduction rate will only be measured for patients undergoing IHIPEC. This rate is defined by the percentage of patients who receive a CC0 (indicates no residual tumor visible to the naked eye) or CC1 (indicates minimal residual tumor visible) after completing the IHIPEC protocol. This metric assesses the ability of MRT-selected personalized IHIPEC to downstage PM tumor burden and improve the rate of resection.
Mean MRT Turnaround Time | up to 12 months
  The mean time in days that it takes for MRT personalized drug readouts to come back to the medical team will be recorded: from the time the biopsy is shipped to Travera to the time the personalized drug readouts are made accessible to the medical team.
MRT Success Rate | up to 12 months
  The percentage of MRT results that come back with specific personalized drug readouts will be recorded. This excludes MRT results that were inconclusive or had an inadequate cancer cell sample or insufficient tumor cell purity to conduct MRT.
MRT Tumor Cell Viability | up to 12 months
  The percentage of MRT results that come back as inconclusive due to inadequate tumor cell viability will be recorded. Cell viability can be defined as the percentage of tumor cells that have sufficient metabolic activity to undergo accurate MRT testing as to not receive an inconclusive result.
MRT Tumor Cell Purity: | up to 12 months
  The percentage of MRT results that come back as inconclusive due to inadequate tumor cell purity will be recorded. Tumor cell purity can be defined as the percentage of biopsies submitted for MRT with a sufficient proportion of malignant cancer cells in the tumor mass as to not receive an inconclusive result.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Turaga, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No